CLINICAL TRIAL: NCT03552224
Title: Evaluation of the Global Auditory Nerve Activity as a New Method of Electrophysiological Exploration of Hearing in Humans - 2
Brief Title: Evaluation of the Global Auditory Nerve Activity for Exploration of Hearing in Humans
Acronym: MELAUDI-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Institute for Neurosciences of Montpellier U1051 (Unknown); Reims University hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 9890
Record Dates: First submitted 2018-05-23; First posted 2018-06-11 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Hearing Loss
Keywords: Evoked auditory nerve activity; Hearing Loss; Tinnitus
MeSH Terms: conditions — Hearing Loss; Tinnitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subjects with no hearing loss (Experimental): Subjects referred for cerebellopontine angle surgery with no hearing loss with recording of auditory nerve activity by contact electrode
  Interventions: Procedure: Recording of auditory nerve activity
- Subjects with hearing loss (Experimental): Subjects referred for cerebellopontine angle surgery with hearing loss with recording of auditory nerve activity by contact electrode
  Interventions: Procedure: Recording of auditory nerve activity

INTERVENTIONS:
Procedure: Recording of auditory nerve activity — near field recording of auditory nerve activity with contact electrode

SUMMARY:
To date, all the electrophysiological methods for auditory testing rely on the measure on synchronous evoked auditory nerve activity. This measure only takes into account the response of the first action potential in every auditory fibber, but provides no information about the neural response during a sustained activity. This can explain why in experimental models, a loss of more of 80% of auditory nerve fibbers cannot be detected by usual electrophysiological measurements. In this study we aim at investigating the global spontaneous and sound evoked auditory nerve activity by recording directly the electrical field by an electrode placed directly on the auditory nerve of subjects during a skull base surgical procedure. We expected to demonstrated differences in the electrical activity between subjects with or without hearing loss.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 80 years ( inclusive borders)
* patient having to undergo surgery at the level of the ponto-cerebellar angle (microvascular decompression, vestibular neurotomy, tumor resection of the meningioma type or schwannoma) and
* Unaffected by neuro-sensory hearing loss, defined by mean auditory thresholds of less than 20 dB in tone audiometry in bone conduction on the side of the ear to be operated (N = 15, Group 1) or
* Showing mild to moderate hearing loss defined by average hearing loss (average of 500, 1000, 2000 and 4000 Hz thresholds) greater than 20 dB and less than 55 dB in air conduction threshold tone audiometry (N = 15 Group 2).
* Voluntary subjects to participate in the study,
* Subjects having signed written consent to participate in the study,
* Easily accessible topics.

Exclusion Criteria:

* Subjects unable to understand the nature and goals of the study and / or having difficulty communicating with the investigator,
* Subjects refusing to participate, subjects whose free and informed consent has not been sought, subjects for which a consent form has not been signed,
* Subjects for whom there is a contraindication to general anesthesia,
* Subjects with a central neurological pathology that can disrupt electrophysiological recordings
* Not affiliated to a French social security scheme or not benefiting from such a scheme,
* Majors protected by law,
* Pregnant women,
* deprived of liberty by judicial or administrative decision,
* Infectious or inflammatory pathology of the middle ear.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2021-06-26 (Actual); Study Completion 2021-06-26 (Actual)

PRIMARY OUTCOMES:
Amplitude of global evoked auditory nerve activity | 36 months
Spectrum of global evoked auditory nerve activity | 36 months

SECONDARY OUTCOMES:
Mesure of peristimulus time responses of evoked auditory nerve activity | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric VENAIL, PU-PH, Principal Investigator — University Hospital, Montpellier
Locations (1):
- CHU Montpellier, Montpellier, France